CLINICAL TRIAL: NCT04465591
Title: Troponin T Fragmentation in the Assessment of Myocardial Injury Study
Brief Title: TROPOnin FRAGMentation in Myocardial Injury Study
Acronym: Tropo-Fragm
Status: Recruiting | Type: Observational
Sponsor: University of Turku (Other)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, University of Turku
Other Study IDs: T29/2020
Record Dates: First submitted 2020-07-07; First posted 2020-07-10 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Acute Myocardial Infarction Type 1; Myocardial Injury
Keywords: Troponin; myocardial injury; myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Heparin plasma:
  * Troponin T control sample
  * Troponin T fragmentation sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myocardial infarction: Recruited patients with STEMI or NSTEMI and elevated Troponin T
  Interventions: Diagnostic Test: troponin T fragmentation test
- Myocardial injury: Recruited patients with myocardial injury based on elevated Troponin T and associated with renal failure, severe infection, strenouos exercise, atrial fibrillation, myocarditis, takotsubo cardiomyopathy or other similar conditions
  Interventions: Diagnostic Test: troponin T fragmentation test

INTERVENTIONS:
Diagnostic Test: troponin T fragmentation test — laboratory test from blood sample

SUMMARY:
Troponin T (TnT) is a part of the troponin protein complex that principally exists in cardiac and skeletal muscle cells and is widely used as diagnostic biomarker for myocardial injury and, thus, myocardial infarction (MI). Elevated TnT levels can, however, be observed in the presence of other clinical conditions such as heart failure, sepsis and kidney failure and the contemporary high-sensitivity TnT test may yield false positive results when performing diagnostics for suspected MI in these patients.

Recent data have demonstrated that in the presence of MI, TnT gradually undergoes fragmentation into smaller fragments. It has been suggested that in the presence of e.g. chronic kidney disease or physical exercise the released TnT is predominantly in the form of smaller fragments.

However, the clinical significance of TnT fragmentation is unknown and, thus, we sought to investigate the prevalence of fragmentation of TnT in different patient cohorts.

DETAILED DESCRIPTION:
Modern cardiac troponin T (cTnT) tests are highly sensitive in diagnosing AMI and myocardial damage. Atrial fibrillation and many non-cardiac conditions and even strenuous exercise are associated with elevated cTnT levels which are problematic to clinicians and may lead to redundant use of diagnostic coronary angiography or "overdiagnosis" of ACS in the emergency room workup.

The cardiac troponin (cTn) complex is part of the thin filaments of myocardium. Small part (approximately 5% of total content) of troponins are cytosolic. These smaller cytosolic fragments may more easily traverse across cell membranes that have become leaky for some reason but not irreversibly damaged. Only cytoplasmic forms of troponin are contained in the subcellular blebs which lyse upon early cTn release into the circulation. Bleb formation may explain how troponin can appear in blood in the absence of cell necrosis. Still many aspects of their intramyocardial degradation, their tissue release, and their degradation within and elimination from the human circulation are still incompletely understood.

In the early hours of AMI, troponin is found in its full-size complex, but the complexed cTnT degrades in a time-dependent pattern after the first hours. Small molecular weight troponin fragments originating from the cytoplasm may traverse across leaky cell membranes not completely damaged in various conditions without irreversible myocardial cell necrosis.

Commercial cTnT test detects all these fragments and may thus lead to false diagnosis of AMI. At present, there is limited information based on small studies using complicated gel filtration chromatography and Western blotting showing cTnT fragmentation in later phases of AMI and in renal failure. These time-consuming analytical methods are, however, not suitable for clinical purposes in the emergency room.

ANALYTICAL METHODS In this study we test a novel sensitive time-resolved immunofluorometric assay, which has been developed at the biotechnology unit of the Department Biochemistry, University of Turku, which enables us to measure cTnT from blood samples in its intact or only slightly fragmented form. Thus, we can exclude the highly fragmented short forms of cTnT from the analysis. This selectivity can be achieved with specific capture and tracer antibodies that bind to carefully chosen epitopes located closer to the opposite ends of the cTnT molecule. In the assay one of the antibodies is attached to a surface and acts as an antigen capturing antibody. The capture-antigen pair can be detected with tracer antibody, thus forming capture-antigen-tracer complex. In our case this tracer antibody has been labeled with europium chelates which provide sensitive detection by time-resolved fluorometry.

The aim of Tropo-Fragment study is to use the described preliminary assay format in the clinical studies to evaluate:

* TnT fragmentation and its time course in STEMI and NSTEMI
* TnT fragmentation in renal failure, sepsis, strenuous exercise, stroke, atrial fibrillation, takotsubo, myocarditis and healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Troponin T fragmentation sample collected from a recruited patient.

Exclusion Criteria:

* Age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are prospectively recruited from the Heart Center, Department of Medicine and Kidney Center of the study hospital. All patients aged 18 years are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-04-02 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The fragmentation rate of Troponin T | Baseline
  The proportion of fragmented Troponin T in patient cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Juhani K Airaksinen, MD, PhD, Principal Investigator — University of Turku
Locations (2):
- Turku University Hospital, Heart Center, Turku, Southwest Finland, Finland
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Aalto R, Lahtinen A, Airaksinen KEJ, Vasankari T, Hellman T, Koskimaki L, Wittfooth S. Design and Analytical Evaluation of an Immunoassay for Long Forms of Cardiac Troponin T. J Appl Lab Med. 2026 Jan 5;11(1):36-47. doi: 10.1093/jalm/jfaf143. PMID 41025697
- [Derived] Airaksinen JKE, Tuominen T, Paana T, Hellman T, Vasankari T, Salonen S, Junes H, Linko-Parvinen A, Pallari HM, Strandberg M, Teppo K, Jaakkola S, Wittfooth S. Novel troponin fragmentation assay to discriminate between Takotsubo syndrome and acute myocardial infarction. Eur Heart J Acute Cardiovasc Care. 2024 Dec 3;13(11):782-788. doi: 10.1093/ehjacc/zuae115. PMID 39422200
- [Derived] Salonen SM, Tuominen TJK, Raiko KIS, Vasankari T, Aalto R, Hellman TA, Lahtinen SE, Soukka T, Airaksinen KEJ, Wittfooth ST. Highly Sensitive Immunoassay for Long Forms of Cardiac Troponin T Using Upconversion Luminescence. Clin Chem. 2024 Aug 1;70(8):1037-1045. doi: 10.1093/clinchem/hvae075. PMID 38888909
- [Derived] Airaksinen KEJ, Aalto R, Hellman T, Vasankari T, Lahtinen A, Wittfooth S. Novel Troponin Fragmentation Assay to Discriminate Between Troponin Elevations in Acute Myocardial Infarction and End-Stage Renal Disease. Circulation. 2022 Nov;146(18):1408-1410. doi: 10.1161/CIRCULATIONAHA.122.060845. Epub 2022 Oct 31. No abstract available. PMID 36315607